CLINICAL TRIAL: NCT02720705
Title: Transbucal Dexmedetomidine for the Prevention of Emergence Agitation After Sevoflurane Anaesthesia in Pre-school Children
Brief Title: Transbucal Dexmedetomidine for Prevention of Sevoflurane Emergence Agitation in Pre-school Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, MD, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AssuitU
Record Dates: First submitted 2016-03-17; First posted 2016-03-28 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Agitation
Keywords: sevoflurane emergence agitation
MeSH Terms: conditions — Psychomotor Agitation | interventions — Dexmedetomidine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DEX I (Active Comparator): active comparator receive 0.5µg/kg dexmedetomidine orally half an hour before operation
  Interventions: Drug: Dexmedetomidine
- Saline Control (Placebo Comparator): 2ml oral 0.9%saline half an hour before operation
  Interventions: Drug: saline
- DEX II (Active Comparator): active comparator receive,1µg/kg dexmedetomidine orally half an hour before operation
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — oral dexmedetomidine
  Other Names: precedex
  Arms: DEX I; DEX II
Drug: saline — 2ml 0.9% saline administered orally half an hour before induction of anesthesia
  Other Names: 0.9% saline
  Arms: Saline Control

SUMMARY:
The aim of this study is to evaluate the efficacy of transbucal dexmedetomidine given in preschool children undergoing tonsillectomy operations in the prevention sevoflurane agitation.

DETAILED DESCRIPTION:
Agitation during the emergence from general anesthesia is a great post-operative problem that often injures the patients themselves and requires the medical staff to restrain and calm them. The predisposing factors for emergence agitation include anesthesia, operation, and patient. Sevoflurane anesthesia results in higher incidence of emergence agitation than halothane, because of the rapid emergence, and its effects on central nervous system inducing convulsion and post-operative behavioral changes. The otorhinolaryngologic and ophthalmologic surgeries, post-operative pain, young age, pre-operative anxiety, no past surgical history, and adjustment disorder of patients are risk factors.

Dexmedetomidine (DEX), a selective α (2)-adrenoreceptor agonist. Intravenous DEX used after induction of anesthesia reduced sevoflurane-associated EA and postoperative pain in pediatric ambulatory surgery.

The investigators designed this study to prove the efficacy of oral dexmedetomidine a selective α (2)-adrenoreceptor agonist, on emergence agitation (EA), recovery profiles, and parents' satisfaction after sevoflurane anesthesia in tonsillectomy.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II patients
* aged 2-6 years
* patient scheduled for elective tonsillectomy due to recurrent
* chronic tonsillitis

Exclusion Criteria:

* patients with known hypersensitivity to medication drugs
* coagulation disorders
* thrombocytopenia
* significant cardiac
* renal
* pulmonary
* hepatic disease

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
The agitation score up to 1hour postoperative. | first postoperative hour
  Agitation intensity will be assessed postoperatively by using agitation score 0= child is asleep. awake/calm =1. irritable/ consolable cry =2. inconsolable cry =3.the child is agitating and thrashing and restlessness Emergence delirium ≥ 3 agitation score will be performed in the following time points; at 5 min postoperative,10 min, 15, 30, 45, 60 min.

SECONDARY OUTCOMES:
Pain score assessed using the objective pain scale. | up to 1hour postoperative hour
  Pain intensity will be assessed postoperatively by using the objective pain scale. objective pain scale assessments will be performed in the following time points; at 5 min postoperative, 10 min, 15, 30, 45, 60 min.

CONTACTS AND LOCATIONS:
Overall Officials: Halla s Abdel-Ghaffar Abdel-Ghaffar, MD, Principal Investigator — assisstant professor in anesthesia and intensive care departement,faculty of medicine,Assiut university,Egypt
Locations (1):
- Assiut university hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdel-Ghaffar HS, Abdel-Wahab AH, Roushdy MM. [Oral trans-mucosal dexmedetomidine for controlling of emergence agitation in children undergoing tonsillectomy: a randomized controlled trial]. Braz J Anesthesiol. 2019 Sep-Oct;69(5):469-476. doi: 10.1016/j.bjan.2019.06.012. Epub 2019 Oct 28. PMID 31672419